CLINICAL TRIAL: NCT03278145
Title: Dependence Receptors in Childhood Acute Leukemia
Brief Title: Dependence Receptors and Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0806
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Genetic Linkage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspiration sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric acute leukemia: Patients of the Institute of Hematology and Pediatric Oncology (IHOPe) with acute leukemia (LA) who came for initial diagnosis, relapse, or at the time of their remission .
  Interventions: Genetic: Genetic analyses

INTERVENTIONS:
Genetic: Genetic analyses — Patients treated at the Institute of Hematology and Pediatric Oncology (IHOPe), a department of Prof. Y. Bertrand, for acute leukemia (LA) at the time of diagnosis initial, or relapse, after obtaining signed parental consent. The same patients will benefit from a new sample at the time of their remission balance. Analyses for this research will be made from bone marrow aspiration samples performed for diagnosis and treatment of these patients. The medical team will investigate whether RDs, in particular DCC, are expressed in acute leukemia cells at the time of diagnosis or relapse and then in these patients at the time of the remission balance. This research will be both qualitative and quantitative. Next, investigators will characterize the existence and then the level of expression of the ligand specific for DCC, Netrin-1, in these same leukemic cells, at the time of diagnosis / relapse and remission.

SUMMARY:
Acute leukaemias (AL) are the first cause of cancer in children, with a majority of B acute lymphoblastic leukemia (ALL). Some of the processes causing leukemogenesis are already identified and well characterized in some AL subtypes such as translocation t (12; 21) of good prognosis in ALL. However, translocations are not sufficient to explain all the different processes of leukemogenesis, and other processes such as genetic / epigenetic mutations leading to oncogene activation / inhibition of tumor suppressor genes are the object research. Among the latter, mutations in tumor suppressor genes such as DCC (Deleted in Colorectal Cancer) have recently been identified in solid cancers, such as in hemopathies. This gene was subsequently characterized as encoding a "dependence receptor" specifically binding to its Netrin-1 ligand.

Dependence receptors (RDs) are transmembrane receptors that cause cell death in the absence of their ligand. RD decreases tumor progression and overexpression of their ligands is observed in many cancers, such as B lymphomatous hemopathies in adults. Inhibition of the RD-ligand interaction constitutes a new and original therapeutic target in oncology.

The aim of this study is to investigate whether RDs, in particular DCC, are expressed in acute leukemia cells at the time of diagnosis or relapse in patients aged 1 to 18 years, and then in these patients at the time of the remission balance. This research will be both qualitative and quantitative.

ELIGIBILITY:
Inclusion Criteria:

* aged between 1 and 18 years
* taken care of at the Institute of Hematology and Pediatric Oncology (Service of Professor Yves Bertrand, IHOPe)
* for acute lymphoblastic or myeloblastic leukemia
* initial diagnosis or relapse
* who do not have a vital emergency criterion at the time of taking care (see exclusion criteria)
* affiliated to a social security scheme (100% assumed)
* after signing the informed consent of the holders of parental authority

Exclusion Criteria:

* less than 1 year, or more than 18 years to diagnosis
* with chronic leukemia
* severe anemia at diagnosis (hemoglobin <40g / l), or a state of shock whatever the cause (infectious, cardiogenic, hypovolemic)

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The target population consists of patients aged 1 to 18 years treated at the Institute of Hematology and Pediatric Oncology (IHOPe), a department of Prof. Y. Bertrand, for acute leukemia (LA) at the time of diagnosis initial, or relapse, after obtaining signed parental consent. The same patients will benefit from a new sample at the time of their remission balance.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Detection of specific labeling of the DCC-dependent receptor on the surface of leukemic cells | Maximum 4 months (sampling at the time of diagnosis / relapse and remission)
  Primary endpoint: presence of specific labeling of the DCC-dependent receptor on the surface of leukemic cells that will be detectable in flow cytometry.
  This marking will be both qualitative (positive signal = presence of the receptor, absence of signal = absence of the receptor), and quantitative (percentage of expression of the receptor on the surface of the cells).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, France

IPD SHARING:
Plan to Share IPD: No